CLINICAL TRIAL: NCT01021111
Title: The Design and Evaluation of an Active Intervention for the Prevention of Non-contact ACL Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Peter Andriacchi, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SU-09242009-4061; 16584 (Other: Stanford University Institutional Review Board)
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Athletic Injuries; Sprains and Strains; Wounds and Injuries; Knee Injuries
MeSH Terms: conditions — Athletic Injuries; Sprains and Strains; Wounds and Injuries; Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Activity Training with Feedback (Experimental): Subject is tested prior to training and retested with feedback training designed to modify the mechanics of landing during jumping and running activities
  Interventions: Device: Activity Training with Feedback

INTERVENTIONS:
Device: Activity Training with Feedback — The feedback system consisted of three small inertial measurement units affixed on the chest, thigh, and shank segment respectively. These units were connected to a computer that recorded the signal from the inertial sensors at 240 Hz during the jump task. Using custom software, the knee flexion angle, trunk lean, and coronal thigh angular velocity were calculated immediately after the subject completed the jump trial. A projector was used to display the results of the jump analysis. It took less than 10 minutes to place this system on a subject and less than five seconds to analyze a jump.

SUMMARY:
The overall goal of this project is to reduce the risk for anterior cruciate ligament injuries by designing a targeted intervention that will alter the known kinematic and kinetic risk factors associated with ACL injuries.

DETAILED DESCRIPTION:
This study will address the following specific aims: 1) To optimize a wearable, targeted, active training feedback device to reduce the risk of ACL injury among healthy subjects by inducing patterns of movement that alter the known kinematic and kinetic risk factors associated with ACL injuries. 2) To evaluate the efficacy of the active device and determine if the device reduces the risk of ACL injury among healthy subjects by effectively inducing patterns of movement that alter the known kinematic and kinetic risk factors associated with ACL injuries.

ELIGIBILITY:
Inclusion Criteria:The ages would range from 18 to 65. Both male and female subjects will be enrolled, and ethnic backgrounds would be mixed. Exclusion Criteria:(i) chronic lower body pain (ii) recent surgery of the lower or upper body (limitation of range of motion) (iii) previous history of ligament, meniscal, or chondral injury requiring surgery to the lower limb (iv) inability to complete jumping tasks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Peter Andriacchi, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were involved in sports involving jumping maneuvers at the recreational level and free of previous lower limb musculoskeletal injuries, surgery, or pain. Subjects were unaware of the goals of the study prior to the start of the testing session.
Groups:
- Activity Training With Feedback: Subject is tested prior to training and retested with feedback training designed to modify the mechanics of landing during jumping and running activities
  Anterior Cruciate Ligament Measurement and Feedback System
Period: Overall Study
Arm/Group | Activity Training With Feedback
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Activity Training With Feedback: Subjects who underwent activity training with feedback
Arm/Group | Activity Training With Feedback
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 17
Knee Flexion Angle [Mean (Standard Deviation); unit: degrees] | 88.8 (8.0)
Trunk lean [Mean (Standard Deviation); unit: degrees] | 23.6 (8.0)
Thigh coronal angular velocity [Mean (Standard Deviation); unit: degrees/second] | 67.7 (49.7)

OUTCOME MEASURES:

1. Primary Outcome: Knee Flexion Angle and Trunk Flexion Angle After Activity Training With Feedback
Description: Knee flexion angle describes the angle between the tibia and femur during the activity. Trunk flexion is the angle between the shoulders and the hips during the activity.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Activity Training With Feedback
Number analyzed (Participants) | 17
degrees
  Knee Flexion Angle | 105.0 (5.6)
  Trunk Lean | 41.0 (3.8)
Statistical Analysis 1: Comparison: Activity Training With Feedback; The values from the three jumps were averaged in order to have one mean value per subject per session. Paired Student t-tests (baseline vs. follow-up) were used to evaluate the effects of the training; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

2. Secondary Outcome: Thigh Coronal Angular Velocity After Feedback Training
Description: How fast the thigh is moving relative to the tibia during the activity, measured in degrees/second.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: degrees/second
Arm/Group | Activity Training With Feedback
Number analyzed (Participants) | 17
degrees/second | 47.6 (40.5)
Statistical Analysis 1: Comparison: Activity Training With Feedback; The association between the change in the thigh coronal angular velocity from baseline to follow-up and the change in the knee abduction moment from baseline to follow-up was assessed with the Pearson correlation coefficient (R), alpha =0.05; Test type: Superiority or Other; p < 0.05, Pearson

ADVERSE EVENTS:
Time Frame: 1 day
Description: Adverse events were monitored on the day of subject testing
Arm/Group | Activity Training With Feedback
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes